CLINICAL TRIAL: NCT05035797
Title: Impact of Cardiopulmonary Rehabilitation on Weaning of Extracorporeal Membrane Oxygenation (CaRe-ECMO): a Prospective Multidisciplinary Randomized Controlled Clinical Trial
Brief Title: CaRe-ECMO Program on ECMO Weaning
Acronym: CaRe-ECMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yu Zheng, Attending doctor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CaRe-ECMO
Record Dates: First submitted 2021-08-26; First posted 2021-09-05 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Critical Illness
Keywords: Extracorporeal Membrane Oxygenation; Cardiopulmonary Rehabilitation; Weaning; Multidisciplinary; Randomized controlled trial; Open-label
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CaRe-ECMO group (Active Comparator): Patients in the CaRe-ECMO group will be treated with usual care, ECMO therapy, and cardiopulmonary rehabilitation program.
  Interventions: Procedure: Cardiopulmonary rehabilitation; Procedure: Usual care
- Control group (Placebo Comparator): Usual care and ECMO therapy
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Cardiopulmonary rehabilitation — Cardiopulmonary rehabilitation program which encompasses six evidence-based components according to literature review: 1) positioning; 2) passive range of motion (PROM) training; 3) neuromuscular electronic stimulation (NMES); 4) surface electrical phrenic nerve stimulation (SEPNS); 5) PNF techniques; and 6) airway clearance techniques; Usual care normally comprises pharmacotherapy, mechanical ventilation, continuous renal replacement therapy (CRRT), intra-aortic balloon pump (IABP), and specific nursing for ECMO therapy and their original injuries, as appropriate.
  Arms: CaRe-ECMO group
Procedure: Usual care — Control group will be treated with usual care and ECMO therapy. Usual care normally comprises pharmacotherapy, mechanical ventilation, continuous renal replacement therapy (CRRT), intra-aortic balloon pump (IABP), and specific nursing for ECMO therapy and their original injuries, as appropriate.

SUMMARY:
Mortality of patients suffering critical illness has been dramatically improved with advanced technological development of extracorporeal membrane oxygenation (ECMO) therapy. However, weaning rate stayed low in a majority of ECMO-supported patients. As one of several options, cardiopulmonary rehabilitation serves as effective intervention in the improvement of cardiovascular and respiratory function in various major critical illness. Nonetheless, its roles in facilitating ECMO weaning has not yet been explored. The purpose of this study is to investigate the effectiveness of cardiopulmonary rehabilitation on rate of ready for weaning in ECMO-supported patients (CaRe-ECMO).

DETAILED DESCRIPTION:
Studies have documented that rate of mechanical ventilation weaning was improved in patients received early rehabilitation intervention while its effectiveness in ECMO weaning remains unclear. This inspires us to hypothesize that if the medical rationale is based on its assumed benefits on cardiac function and oxygenation, then cardiopulmonary rehabilitation may subsequently contribute to earlier weaning of ECMO. The "CaRe-ECMO" trial is a prospective, multidisciplinary, randomized controlled, parallel group, clinical trial. Cardiopulmonary rehabilitation program which encompasses six evidence-based components:1) positioning; 2) passive range of motion (PROM) training; 3) neuromuscular electronic stimulation (NMES); 4) surface electrical phrenic nerve stimulation (SEPNS); 5) respiratory PNF techniques 6) airway clearance techniques; 366 ECMO-supported patients in department of emergency medicine will be randomized to control and CaRe-ECMO group. CaRe-ECMO group will be treated with usual care, ECMO therapy, and cardiopulmonary rehabilitation program. Usual care normally comprises pharmacotherapy, mechanical ventilation, continuous renal replacement therapy (CRRT), intra-aortic balloon pump (IABP), and specific nursing for ECMO therapy and their original injuries, as appropriate. Control group will be treated with usual care, ECMO therapy. The primary objective of the CaRe-ECMO trial is to investigate the impact of cardiopulmonary rehabilitation combined with usual care on rate of ready for ECMO weaning at CaRe-ECMO Day 7, when compared to usual care alone. Secondary objectives are to evaluate the effects of cardiopulmonary rehabilitation on rate of ECMO weaning, total length of ready for ECMO weaning, total length of ECMO weaning, rate of mechanical ventilation weaning, total length of mechanical ventilation, all-cause mortality, rate of major post-ECMO complications, diaphragmatic thickness and mobility, ECMO Unit length of stay (LOS), total hospital LOS, total cost for hospitalization, cerebral performance category (CPC) index, activity of daily living (ADL), and health related quality of life (HRQoL). The CaRe-ECMO trial is designed to test the hypothesis that early cardiopulmonary rehabilitation can accelerate weaning of ECMO-supported patients. If CaRe-ECMO trial results in superior improvement in primary and secondary outcomes, it will offer an innovative treatment option for ECMO-supported patients.

ELIGIBILITY:
Inclusion Criteria:

1) Aged 18yr or order 2) Eligible for receiving ECMO (veno-venous [VV] or veno-arterial [VA]) therapy 3) With mechanical ventilation 4) With stable condition and eligible for cardiopulmonary rehabilitation after 72 hours of ECMO 5) With no contraindications for cardiopulmonary rehabilitation 6) With a life expectancy of more than 3 days 7) Sign informed consent form by the guardian

Exclusion Criteria:

1) Pregnant 2) Use ECMO as a bridge to recovery or definitive treatment (e.g. lung transplantation or heart transplantation) 3) Enrolled in another trial previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of ready for ECMO weaning at CaRe-ECMO Day 7 | CaRe-ECMO Day 7
  Rate of ready for ECMO weaning will be calculated 7 days after cardiopulmonary rehabilitation delivery

SECONDARY OUTCOMES:
Rate of ready for ECMO weaning | CaRe-ECMO Day 14, 30 and 90
  Rate of ready for ECMO weaning will be calculated 14, 30 and 90 days after cardiopulmonary rehabilitation delivery
Rate of ECMO weaning | CaRe-ECMO Day 7, 14, 30 and 90
  Rate of ECMO weaning will be calculated according to date of ECMO weaning fulfilled
Total length of ready for ECMO weaning | From date of ECMO initiation until the date of ready for ECMO weaning, assessed up to CaRe-ECMO Day 90
  Total length of ready for ECMO weaning refers to exact length in day till patients fulfill all criteria of ready for ECMO weaning according to daily checkout records
Total length of ECMO weaning | From date of ECMO initiation until the date of ECMO weaning, assessed up to CaRe-ECMO Day 90
  Total length of ECMO weaning refers to exact length in day for patients treated with ECMO therapy
Rate of mechanical ventilation weaning | CaRe-ECMO Day 7, 14, 30 and 90
  Rate of mechanical ventilation weaning will be calculated according to date of mechanical ventilation weaning fulfilled. Daily screening of mechanical ventilation weaning will be strictly performed with checklist
Total length of mechanical ventilation | From date of mechanical ventilation initiation until the date of mechanical ventilation weaning, assessed up to CaRe-ECMO Day 90
  Total length of mechanical ventilation refers to exact length in day for patients treated with mechanical ventilation
All-cause mortality | CaRe-ECMO Day 7, 14, 30 and 90
  All-cause mortality is defined as rate of death due to any causes and will be calculated according to date of death
Major complications | CaRe-ECMO Day 7, 14, 30 and 90
  Rate of complications occurred after ECMO, including but not limited to ECMO related complications (e.g., thromboembolism), mechanical ventilation related complications (e.g., pneumonia), newly developed myocardial infarction, acute kidney injury, neurologic events (e.g., stroke, seizures), and multiple organ failure
Diaphragmatic thickness and mobility | Every three days, assessed up to CaRe-ECMO Day 90
  Diaphragmatic thickness and mobility refer to ultrasound guided evaluation of diaphragmatic thickness and mobility under M mode
ECMO Unit length of stay (LOS) | Discharge day (discharge from ECMO Unit), assessed up to CaRe-ECMO Day 90
  ECMO Unit length of stay (LOS) accounts for length in day for patients' stay in the ECMO Unit
Total hospital length of stay | Discharge day (discharge from hospital), assessed up to CaRe-ECMO Day 90
  Total hospital LOS accounts for total hospital LOS in day for patients' stay in both ECMO Unit and other departments
Total cost for hospitalization | Discharge day (discharge from hospital), assessed up to CaRe-ECMO Day 90
  Total cost for hospitalization will be calculated by addition of the cost of all units and departments admission
Cerebral performance category (CPC) index | CaRe-ECMO Day 7, 14, 30, 90 and discharge day (discharge from ECMO Unit), assessed up to CaRe-ECMO Day 90
  Cerebral performance category (CPC) index will be recorded, for those successfully weaning of ECMO, to reflect post-ECMO neurological status
Activity of daily living (ADL) | CaRe-ECMO Day 7, 14, 30, 90 and discharge day (discharge from ECMO Unit), assessed up to CaRe-ECMO Day 90
  Activity of daily living (ADL) will be evaluated, for those successfully weaning of ECMO, with Katz Index
Health related quality of life (HRQoL) | CaRe-ECMO Day 7, 14, 30, 90 and discharge day (discharge from ECMO Unit), assessed up to CaRe-ECMO Day 90
  Health related quality of life (HRQoL) will be measured, for those successfully weaning of ECMO, with SF-12

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Lu, M.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Jingsong Zhang, M.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Xufeng Chen, M.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No